CLINICAL TRIAL: NCT00699582
Title: A Double-Blind, Placebo-Controlled, Dose-Escalation, Parallel-Group Study to Evaluate the Efficacy and Safety of E2007 (Perampanel) Given as Adjunctive Therapy in Subjects With Refractory Partial Seizures
Brief Title: To Evaluate The Efficacy and Safety of E2007 (Perampanel) Given as Adjunctive Therapy in Subjects With Refractory Partial Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2007-G000-305; 2007-006168-31 (EudraCT Number)
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Results first posted 2012-11-22 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2012-10

CONDITIONS: Refractory Partial Seizures
Keywords: E2007 (perampanel); refractory partial seizures; adjunctive therapy; seizure frequency; reduction in seizure frequency; partial onset seizures; safety; concomitant AED(s)
MeSH Terms: conditions — Seizures | interventions — perampanel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: E2007 (perampanel)
- 2 (Experimental)
  Interventions: Drug: E2007 (perampanel)
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E2007 (perampanel) — 8 mg perampanel in a 1:1:1 ratio, 125 subjects/arm. All subjects will take a maximum of 6 tablets daily for the duration of the study and will be up-titrated weekly in 2-mg increments to their randomized dose.
  Other Names: perampanel
  Arms: 1
Drug: E2007 (perampanel) — 12 mg perampanel in a 1:1:1 ratio, 125 subjects/arm. All subjects will take a maximum of 6 tablets daily for the duration of the study and will be up-titrated weekly in 2-mg increments to their randomized dose.
  Other Names: perampanel
  Arms: 2
Drug: Placebo — Placebo in a 1:1:1 ratio, 125 subjects/arm. All subjects will take a maximum of 6 tablets daily for the duration of the study.
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of perampanel when given as an adjunctive therapy in subjects with refractory partial seizures.

ELIGIBILITY:
Inclusion criteria:

Each subject must meet all of the following criteria to be enrolled in this study:

1. Provide written informed consent signed by the subject or legal guardian prior to entering the study or undergoing any study procedures (If the written informed consent is provided by the legal guardian because the subject is unable to do so, a written or verbal assent from the subject must also be obtained).
2. Be considered reliable and willing to be available for the study period and able to record seizures and report Adverse Events (AEs) them self or have a caregiver who can record seizures and report AEs for them.
3. Male or female and greater than or equal to 12 years of age (within the course of the study), or greater than or equal to 18 years of age (depending on location) at the time of signing the informed consent.
4. Females should be either of non-childbearing potential (defined as having undergone surgical sterilization, or postmenopausal [age 50 and amenorrheic for 12 months]) or of childbearing potential. Females of childbearing potential must have a negative serum beta-human chorionic gonadotropin (ß-hCG) at Visit 1 and a negative urine pregnancy test prior to randomization at Visit 2. Female subjects of childbearing potential must agree to be abstinent or to use at least 1 medically acceptable method of contraception (eg, a double-barrier method [eg, condom + spermicide, condom + diaphragm with spermicide], IUD, or have a vasectomised partner) starting at Visit 1 and throughout the entire study period and for 2 months after the last dose of study drug. Those women using hormonal contraceptives must also be using an additional approved method of contraception (as described previously) starting at Visit 1 and continuing throughout the entire study period and for 2 months after the last dose of study drug. (It is not required for male subjects to use contraceptive measures based on preclinical toxicology data).
5. Have a diagnosis of epilepsy with partial seizures with or without secondarily generalized seizures according to the International League Against Epilepsy's Classification of Epileptic Seizures (1981). Diagnosis should have been established by clinical history and an electroencephalogram (EEG) that is consistent with localization-related epilepsy; normal interictal EEGs will be allowed provided that the subject meets the other diagnosis criterion (ie, clinical history).
6. Have had a computed tomography (CT) or magnetic resonance imaging (MRI) within the last 10 years that ruled out a progressive cause of epilepsy.
7. Have uncontrolled partial seizures despite having been treated with at least 2 different anti-epileptic drugs (AEDs) within approximately the last 2 years.
8. During the 6-week Pre-randomization Phase subjects must have had ≥5 partial seizures (with ≥2 partial seizures per each of 3-week period) and with no 25-day seizure-free period in the 6-week period, as documented via a valid seizure diary. Only simple partial seizures with motor signs, complex partial seizures, and complex partial seizures with secondary generalization are counted toward this inclusion.
9. Are currently being treated with stable doses of 1, 2 or a maximum of 3 approved AEDs. Only 1 inducer AED (defined as; carbamazepine, phenytoin, phenobarbital, or primidone only) out of the maximum of 3 AEDs is allowed.
10. Are on a stable dose of the same concomitant AED(s) for 1 month (or no less than 21 days) prior to Visit 1; in the case where a new AED regime has been initiated for a subject, the dose must be stable for 2 months (or no less than 49 days) prior to Visit 1.
11. If on a stable dose (other than intermittent rescue use) of benzodiazepines for epilepsy (or for anxiety or sleep disorders) the prescribed dose must be stable for 1 month (or no less than 21 days) prior to Visit 1. (Note: the use of intermittent rescue benzodiazepines is defined in the exclusion criterion #22 below.) When used in these cases (epilepsy, anxiety or sleep disorders), benzodiazepines will be counted as 1 AED; therefore, only 1 or a maximum of 2 additional approved AEDs will be allowed.
12. A vagal nerve stimulator (VNS) is allowed but it must have been implanted ≥5 months prior to Visit 1. Stimulator parameters can not be changed for 1 month (or no less than 21 days) prior to Visit 1 or thereafter during the study.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. Participated in a study involving administration of an investigational compound or device within 1 month (or no less than 21 days) prior to Visit 1, or within approximately 5 half-lives of the previous investigational compound, whichever is longer.
2. Pregnant and/or lactating.
3. Participated in previous perampanel studies.
4. Presence of nonmotor simple partial seizures only.
5. Presence of primary generalized epilepsies or seizures, such as absences and or myoclonic epilepsies.
6. Presence or previous history of Lennox-Gastaut syndrome.
7. A history of status epilepticus within approximately 12 months prior to Visit 1.
8. Seizure clusters where individual seizures cannot be counted.
9. A history of psychogenic seizures.
10. Evidence of clinically significant disease (eg, cardiac, respiratory, gastrointestinal, renal disease) that in the opinion of the Investigator(s) could affect the subject's safety or the study conduct.
11. Scheduled and/or confirmed to have epilepsy surgery within 6 months after Visit 1; however those who have previously documented "failed" epilepsy surgery will be allowed.
12. Evidence of significant active hepatic disease. Stable elevations of liver enzymes, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) due to concomitant medication(s) will be allowed if they are less than 3 times the upper limit of normal (ULN).
13. Evidence of significant active hematological disease; white blood cell (WBC) count <= 2500/µL (2.50 1E+09/L) or an absolute neutrophil count <= 1000/µL (1.00 1E+09/L).
14. A clinically significant ECG abnormality, including prolonged QTc defined as >450 msec.
15. Suffering from psychotic disorder(s) and/or unstable recurrent affective disorder(s) evident by use of antipsychotics or have had a suicide attempt(s) within approximately the last 2 years.
16. Presence of a progressive central nervous system (CNS) disease, including degenerative CNS diseases and progressive tumors.
17. History of drug or alcohol dependency or abuse within approximately the last 2 years.
18. Have had multiple drug allergies or a severe drug reaction to an AED(s), including dermatological (eg, Stevens-Johnson syndrome), hematological, or organ toxicity reactions.
19. If felbamate is used as a concomitant AED, subjects must be on felbamate for at least 2 years, with a stable dose for 2 months (or no less than 49 days) prior to Visit 1. They must not have a history of white blood cell (WBC) count below 2500/µL (2.50 1E+09/L), platelets below 100,000, liver function tests (LFTs) above 3 times the upper limit of normal (ULN), or other indication of hepatic or bone marrow dysfunction while receiving felbamate. If subjects received felbamate in the past, it must have been discontinued 2 months (or no less than 49 days) prior to Visit 1.
20. Concomitant use of vigabatrin. Subjects who took vigabatrin in the past must be off vigabatrin for approximately 5 months prior to Visit 1 and must have documentation showing no evidence of a vigabatrin associated clinically significant abnormality in a visual perimetry test.
21. Concomitant use of barbiturates (except for seizure control indication) within 1 month (or no less than 21 days) prior to Visit 1.
22. Use of intermittent rescue benzodiazepines (ie, 1-2 doses over a 24-hr period considered one-time rescue) 2 or more times in a 1-month period prior to Visit 1; or
23. Any condition(s) that will make the subject, in the opinion of the Investigator, unsuitable for the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2008-05; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Squillacote, M.D., Study Director — Eisai Inc.
Locations (88):
- United States (32):
  - North Alabama Neuroscience Research Associates, Huntsville, Alabama
  - Huntsville, Alabama
  - Xenoscience, Inc., Phoenix, Arizona
  - Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Tucson, Arizona
  - Fresno, California
  - Sacramento, California
  - Neurosearch II, Inc., Ventura, California
  - Ventura, California
  - Mile High Research Center, Denver, Colorado
  - Neurology Associates of Northern Colorado, Fort Collins, Colorado
  - Fort Collins, Colorado
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - Jacksonville, Florida
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - Neurological Research Center at Hattiesburg Clinic, Hattiesburg, Mississippi
  - Hattiesburg, Mississippi
  - The Comprehensive Care Center for Children And Adults, Chesterfield, Missouri
  - Chesterfield, Missouri
  - Saint Luke's Comprehensive Epilepsy Center, Kansas City, Missouri
  - Kansas City, Missouri
  - Buffalo, New York
  - NYU Comprehensive Epilepsy Center, New York, New York
  - New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Syracuse, New York
  - Dallas, Texas
  - Salt Lake City, Utah
  - Dean Foundation for Health, Research and Education, Inc., Madison, Wisconsin
  - Madison, Wisconsin
- Austria (4):
  - Graz
  - Innsbruck
  - Linz
  - Vienna
- Belgium (4):
  - Brussels
  - Ghent
  - Leuven
  - Ottignies (lln)
- Vantaa, Finland
- France (7):
  - Angers
  - Béthune
  - Bron
  - Dijon
  - Montpellier
  - Rennes
  - Toulouse
- Germany (7):
  - Bad Berka
  - Berlin
  - Bernau
  - Bielefeld
  - Bonn
  - Erlangen
  - Göttingen
- India (4):
  - Mangalore, Karnataka
  - Nagpur, Maharashtra
  - Nashik, Maharashtra
  - New Delhi
- Israel (6):
  - Ashkelon
  - Haifa
  - Holon
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
- Italy (3):
  - Florence
  - Milan
  - Napoli
- Netherlands (5):
  - Haarlem
  - Heeze
  - Nijmegen
  - The Hague
  - Zwolle
- Russia (3):
  - Kazan'
  - Moscow
  - Nizhny Novgorod
- South Africa (5):
  - Rosebank, Gauteng
  - Richards Bay, KwaZulu-Natal
  - Cape Town, Western Cape
  - Cape Town
  - Johannesburg
- Sweden (2):
  - Gothenburg
  - Linköping
- United Kingdom (5):
  - Bristol
  - Liverpool
  - London
  - Middlesbrough
  - Stoke-on-Trent

REFERENCES:
- [Derived] Bresnahan R, Hill RA, Wang J. Perampanel add-on for drug-resistant focal epilepsy. Cochrane Database Syst Rev. 2023 Apr 14;4(4):CD010961. doi: 10.1002/14651858.CD010961.pub2. PMID 37059702
- [Derived] Maguire M. Response to "Perampanel and pregnancy: Could experience be a gloomy lantern that does not even illuminate its bearer?". Epilepsy Behav. 2022 Apr;129:108654. doi: 10.1016/j.yebeh.2022.108654. Epub 2022 Mar 16. No abstract available. PMID 35305920
- [Derived] French JA, Gil-Nagel A, Malerba S, Kramer L, Kumar D, Bagiella E. Time to prerandomization monthly seizure count in perampanel trials: A novel epilepsy endpoint. Neurology. 2015 May 19;84(20):2014-20. doi: 10.1212/WNL.0000000000001585. Epub 2015 Apr 15. PMID 25878175
- [Derived] Rosenfeld W, Conry J, Lagae L, Rozentals G, Yang H, Fain R, Williams B, Kumar D, Zhu J, Laurenza A. Efficacy and safety of perampanel in adolescent patients with drug-resistant partial seizures in three double-blind, placebo-controlled, phase III randomized clinical studies and a combined extension study. Eur J Paediatr Neurol. 2015 Jul;19(4):435-45. doi: 10.1016/j.ejpn.2015.02.008. Epub 2015 Mar 5. PMID 25823975
- [Derived] Steinhoff BJ, Ben-Menachem E, Ryvlin P, Shorvon S, Kramer L, Satlin A, Squillacote D, Yang H, Zhu J, Laurenza A. Efficacy and safety of adjunctive perampanel for the treatment of refractory partial seizures: a pooled analysis of three phase III studies. Epilepsia. 2013 Aug;54(8):1481-9. doi: 10.1111/epi.12212. Epub 2013 May 10. PMID 23663001
- [Derived] French JA, Krauss GL, Steinhoff BJ, Squillacote D, Yang H, Kumar D, Laurenza A. Evaluation of adjunctive perampanel in patients with refractory partial-onset seizures: results of randomized global phase III study 305. Epilepsia. 2013 Jan;54(1):117-25. doi: 10.1111/j.1528-1167.2012.03638.x. Epub 2012 Aug 20. PMID 22905857

RESULTS

PARTICIPANT FLOW:
Groups:
- Perampanel 8mg: Perampanel 8mg maximum daily dose (Titration from 2mg to 8mg daily over 6-weeks; Maintenance at 8mg daily over 13-weeks)
- Perampanel 12mg: Perampanel 12mg maximum daily dose (Titration from 2mg to 12mg daily over 6-weeks; Maintenance at 12mg daily over 13-weeks)
Period: Overall Study
Arm/Group | Placebo | Perampanel 8mg | Perampanel 12mg
Started | 138 | 130 | 121
Completed | 120 | 108 | 93
Not Completed | 18 | 22 | 28
Not completed — Adverse Event | 4 | 11 | 23
Not completed — Withdrawal by Subject | 6 | 7 | 4
Not completed — Lack of Efficacy | 1 | 0 | 1
Not completed — Progressive Disease | 1 | 0 | 0
Not completed — Administrative/Other | 4 | 3 | 0
Not completed — Randomized, Not Treated | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Perampanel 8mg | Perampanel 12mg | Total
Number analyzed (Participants) | 138 | 130 | 121 | 389
Age, Customized [Number; unit: participants]
  <18 years | 17 | 17 | 10 | 44
  18-64 years | 120 | 110 | 109 | 339
  >64 years | 1 | 3 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants] — For the placebo arm, there were 2 subjects who were randomized, but not treated. For the perampanel 8mg arm, there was 1 subject who was randomized, but not treated.
  Participants
    Female | 66 | 64 | 71 | 201
    Male | 72 | 66 | 50 | 188
Race/Ethnicity, Customized [Number; unit: participants] — Race
  participants
    White | 117 | 108 | 100 | 325
    Black or African American | 1 | 2 | 1 | 4
    Asian | 12 | 14 | 16 | 42
    American Indian or Alaska Native | 1 | 0 | 0 | 1
    Other | 7 | 6 | 4 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in the 28-day Seizure Frequency From Baseline to the End of the Double-blind Phase (Titration and Maintenance Phases)
Description: Seizure frequency per 28 days was derived from the information recorded in the subject diaries.
Time Frame: Baseline (Pre-randomization) through Week 19
Population: Full Intent-to-Treat (ITT) Analysis Set - group of subjects who were randomized to study drug, received study drug, and had any seizure frequency data during the Doubleblind Phase. For Placebo arm, 2 subjects were randomized but not treated. For Perampanel 8mg arm, 1 subject was randomized but not treated.
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Placebo | Perampanel 8mg | Perampanel 12mg
Number analyzed (Participants) | 136 | 129 | 121
Percent Change | -9.72 [-91.8 to 404.3] | -30.52 [-94.0 to 234.3] | -17.57 [-100.0 to 858.3]

2. Secondary Outcome: Responder Rate
Description: The responder rate for the Full ITT Analysis Set from the maintenance LOCF (Last Observation Carried Forward). A responder was a subject who had a 50 percent or greater reduction in seizure frequency per 28 days from the Pre-randomization phase.
Time Frame: Baseline (Pre-randomization) through Week 19
Population: Full ITT Analysis Set. For Placebo arm, 2 subjects were randomized but not treated. For Perampanel 8mg arm, 1 subject was randomized but not treated.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Perampanel 8mg | Perampanel 12mg
Number analyzed (Participants) | 136 | 129 | 121
Percentage of Participants
  Responders (Yes) | 14.7 | 33.3 | 33.9
  Non-Responders(No) | 85.3 | 66.7 | 66.1

3. Secondary Outcome: Percent Change in the 28-day Complex Partial Plus Secondarily Generalized Seizure Frequency From Baseline to the End of the Double-blind Phase (Titration and Maintenance Phases)
Description: Percent Change in the Seizure frequency per 28 days was derived from the information recorded in the subject diaries.
Time Frame: Baseline (Pre-randomization) through Week 19
Population: Full ITT Analysis Set with Complex Partial plus Secondarily Generalized Seizures at Pre-randomization. For Placebo arm, 2 subjects were randomized but not treated. For Perampanel 8mg arm, 1 subject was randomized but not treated.
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Placebo | Perampanel 8mg | Perampanel 12mg
Number analyzed (Participants) | 126 | 119 | 113
Percent Change | -8.05 [-100.0 to 382.4] | -32.72 [-100.0 to 1023.2] | -21.89 [-100.0 to 733.3]

ADVERSE EVENTS:
Time Frame: From the time the subject signed the informed consent form to 30 days after the last dose of the study drug.
Description: Adverse events (AE) were assessed at clinical visits based on the subject's diary, vitals, weight, physical examination, neurological exam, and laboratory evaluations; and by telephone interviews/contact.
Arm/Group | Placebo | Perampanel 8mg | Perampanel 12mg
Serious Adverse Events (participants affected / at risk) | 7/136 | 10/129 | 12/121
Other Adverse Events (participants affected / at risk) | 55/136 | 90/129 | 90/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=136) | Perampanel 8mg (N=129) | Perampanel 12mg (N=121)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Partial seizures with secondary generalisation (Nervous system disorders) | 0 | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 1
Belligerence (Psychiatric disorders) | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0
Conversion disorder (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Ovarian mass (Reproductive system and breast disorders) | 0 | 0 | 1
Ovarian rupture (Reproductive system and breast disorders) | 0 | 0 | 1
Polycystic ovaries (Reproductive system and breast disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=136) | Perampanel 8mg (N=129) | Perampanel 12mg (N=121)
Constipation (Gastrointestinal disorders) | 4 | 4 | 7
Nausea (Gastrointestinal disorders) | 5 | 11 | 12
Fatigue (General disorders) | 11 | 17 | 20
Irritability (General disorders) | 5 | 12 | 11
Nasopharyngitis (Infections and infestations) | 9 | 10 | 5
Upper respiratory tract infection (Infections and infestations) | 5 | 9 | 5
Fall (Injury, poisoning and procedural complications) | 4 | 6 | 9
Weight Increased (Investigations) | 3 | 7 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 7
Balance Disorder (Nervous system disorders) | 1 | 7 | 3
Convulsion (Nervous system disorders) | 7 | 3 | 5
Dizziness (Nervous system disorders) | 10 | 41 | 58
Headache (Nervous system disorders) | 17 | 11 | 15
Somnolence (Nervous system disorders) | 4 | 16 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No